CLINICAL TRIAL: NCT06658002
Title: Fungal Ulcer Treatment Augmented With Natamycin and Cyclosporine A
Acronym: FANCY
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: Aravind Eye Hospitals, India (Other); Aravind Eye Care System (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 24-41971
Record Dates: First submitted 2024-10-23; First posted 2024-10-26 (Actual); Last update posted 2025-10-06 (Actual); Status verified 2025-10

CONDITIONS: Fungal Keratitis; Corneal Ulcer
Keywords: Corneal Ulcer; Cyclosporine A; Fungal Keratitis; Fungal Corneal Ulcer
MeSH Terms: conditions — Corneal Ulcer | interventions — Cyclosporine

STUDY DESIGN:
Intervention Model Description: This is a randomized controlled trial in which participants with smear or culture proven fungal keratitis are treated for a minimum of 48 hours with topical natamycin and then randomized in a 1:1:1 ratio to receive either topical Cyclosporine A (CsA) 0.1% or CsA 2% or placebo for 4 weeks. In cases of bilateral fungal keratitis, if both eyes fit inclusion criteria, the eye with worse acuity will be randomized.
  The primary outcome is Best Corrected Visual Acuity (BCVA) at 3 months.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The treating and examining doctors and all participants will be masked to the identity of the medication in each group. The study drug will be labeled A, B ,C D, E, F with two letters to each treatment group. The only people who will not be masked is the pharmacist at Pondicherry who relabels the medications with the study drug code and maintains the master key of which drug belongs to which study label, the data analyst responsible for generating the randomization code, and a United States study coordinator who is responsible for relabeling protocol and training. The study coordinator at Aravind will not be informed of the master key but will be aware of the study drug allocation name as he/she will be dispensing study drug to the participant. The study coordinator at Aravind will review the drops with the patient each visit. The participants will be informed to not show the examining doctor any of the medications. The study doctors will not ask to see the study medications.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Cyclosporine A (CsA) 0.1% (Experimental): After one week of hourly natamycin eye drops the participants in this arm will use this drop four times a day for one month then twice a day for one month.
  Interventions: Drug: Cyclosporine A
- Cyclosporine A (CsA) 2% (Experimental): After one week of hourly natamycin eye drops the participants in this arm will use this drop four times a day for one month then twice a day for one month.
  Interventions: Drug: Cyclosporine A
- Placebo (Placebo Comparator): After one week of hourly natamycin eye drops the participants in this arm will use this drop four times a day for one month then twice a day for one month.
  Interventions: Other: Placebo Comparator: Placebo

INTERVENTIONS:
Drug: Cyclosporine A — Participants with smear or culture proven fungal keratitis are treated for a minimum of 48 hours with topical natamycin and then randomized in a 1:1:1 ratio to receive either topical Cyclosporine A (CsA) 0.1%, 2% or placebo for 4 weeks. Natamycin is continued until the ulcer has healed.
  Arms: Cyclosporine A (CsA) 0.1%; Cyclosporine A (CsA) 2%
Other: Placebo Comparator: Placebo — Participants with smear or culture proven fungal keratitis are treated for a minimum of 48 hours with topical natamycin and then randomized in a 1:1:1 ratio to receive either topical Cyclosporine A (CsA) 0.1%, 2% or placebo for 4 weeks. Natamycin is continued until the ulcer has healed.
  Arms: Placebo

SUMMARY:
The goal of this clinical trial is to learn if adjunctive topical Cyclosporine A eye drops combined with standard of care topical Natamycin treatment improves vision outcomes in patients with fungal keratitis.

DETAILED DESCRIPTION:
This is a randomized, masked, clinical trial of patients with documented fungal infections of the cornea. In this trial participants are treated with (standard of care) topical natamycin for a minimum of 48 hours and then randomized in a 1:1:1 ratio to receive either topical Cyclosporine A (CsA) 0.1%, or CsA 2%, or placebo for 4 weeks. Natamycin will be continued until the corneal ulcer has resolved. The primary outcome of this pilot trial is best corrected visual acuity (BCVA) at 3 months. The specific aims of this trial are to:

* to determine if early use of topical cyclosporine A is a beneficial adjuvant to natamycin in the treatment of mild to moderate fungal keratitis.
* to determine if adjunctive 2% cyclosporine A demonstrates greater efficacy than 0.1% cyclosporine A in the treatment of fungal keratitis.
* to determine which ulcer characteristics, predict the most benefit from the addition of early topical cyclosporine.

In this study the investigators will partner with their cornea colleagues at the Aravind Eye Hospital. This is because the incidence of fungal corneal ulcers is among the highest in the world in this location.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion is based on presenting acuity, not ulcer size.
* Inclusion of 20/40 = 6/12 = 0.3 Log MAR and 20/400 = 3/60 = +1.3 Log MAR.
* Smear or culture positive for fungal keratitis, any length.
* Age 18 years.
* Willing to participate in study.

Exclusion Criteria:

* Co-infection with bacterial or viral keratitis.
* Corneal perforation.
* Requiring therapeutic keratoplasty for fungal keratitis.
* Unwilling or unable to follow up (e.g., living too far from hospital).
* Presenting acuity better than 20/40 = 6/12 = 0.3 Log MAR or worse than 20/400 = 3/60 = +1.3 Log MAR.
* Subjects taking cyclosporine at any concentration on presentation.
* Acuity worse than 20/200 = 6/60 = +1.0 Log MAR in unaffected eye.
* Pregnant women.
* Penetrating Keratoplasty.
* Presents with a 0-7 day history of topical steroid.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2025-09-01 (Actual); Primary Completion 2027-09-01 (Estimated); Study Completion 2027-09-01 (Estimated)

PRIMARY OUTCOMES:
Best Corrected Visual Acuity (BCVA) | 3 months (12 weeks)

CONTACTS AND LOCATIONS:
Overall Officials: Gerami D Seitzman, MD, Principal Investigator — UCSF Proctor Foundation
Locations (2):
- University of California, San Farncisco, San Francisco, California, United States
- Aravind Eye Institute, Pondicherry, Tamil Nadu, India

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chatterjee S, Agrawal D. Use of Topical Cyclosporine 0.1% in Therapeutic Penetrating Keratoplasty for Fungal Keratitis. Cornea. 2022 Sep 1;41(9):1116-1121. doi: 10.1097/ICO.0000000000002827. Epub 2021 Sep 3. PMID 34483271
- [Background] Kauss Hornecker M, Charles Weber S, Brandely Piat ML, Darrodes M, Jomaa K, Chast F. [Cyclosporine eye drops: A 4-year retrospective study (2009-2013)]. J Fr Ophtalmol. 2015 Oct;38(8):700-8. doi: 10.1016/j.jfo.2015.02.008. Epub 2015 Sep 11. French. PMID 26371985
- [Background] Bell NP, Karp CL, Alfonso EC, Schiffman J, Miller D. Effects of methylprednisolone and cyclosporine A on fungal growth in vitro. Cornea. 1999 May;18(3):306-13. doi: 10.1097/00003226-199905000-00012. PMID 10336034
- [Background] Perry HD, Doshi SJ, Donnenfeld ED, Bai GS. Topical cyclosporin A in the management of therapeutic keratoplasty for mycotic keratitis. Cornea. 2002 Mar;21(2):161-3. doi: 10.1097/00003226-200203000-00006. PMID 11862086
- [Background] Cordeiro RA, Macedo RB, Teixeira CEC, Marques FJF, Bandeira TJPG, Moreira JLB, Brilhante RSN, Rocha MFG, Sidrim JJC. The calcineurin inhibitor cyclosporin A exhibits synergism with antifungals against Candida parapsilosis species complex. J Med Microbiol. 2014 Jul;63(Pt 7):936-944. doi: 10.1099/jmm.0.073478-0. Epub 2014 Apr 10. PMID 24722799
- [Background] Survase SA, Kagliwal LD, Annapure US, Singhal RS. Cyclosporin A--a review on fermentative production, downstream processing and pharmacological applications. Biotechnol Adv. 2011 Jul-Aug;29(4):418-35. doi: 10.1016/j.biotechadv.2011.03.004. Epub 2011 Apr 5. PMID 21447377